CLINICAL TRIAL: NCT03561389
Title: iFR-guided Revascularization of Non-culprit Lesion in Patients With ST-segment Elevation Myocardial Infarction and Multivessel Disease (WAVE Registry): Long-term Outcome.
Brief Title: iFR-guided Revascularization in STEMI
Acronym: WAVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Principal Investigator, Carmine Musto, Carmine Musto, MD, Principal Investigator, Interventional Cardiology Unit, Azienda Ospedaliera San Camillo Forlanini
Other Study IDs: 76/2018 CE Lazio1
Record Dates: First submitted 2018-05-27; First posted 2018-06-19 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional assessment of non-culprit lesions during percutaneous coronary intervention (PCI) in patients with acute coronary syndrome could improve risk stratification and long-term prognosis. It was previously demonstrated the diagnostic accuracy of instantaneous wave-free ratio (iFR) in functional assessment of non-culprit lesions in multivessel patients with ST-segment elevation myocardial infarction (STEMI), also highlighting the intralesional reproducibility of both fractional flow reserve (FFR) and iFR between baseline and staged. In this study the investigators aimed to verify the clinical impact on long-term outcome of iFR assessment in the acute multivessel setting.

DETAILED DESCRIPTION:
Background - Approximately 40-50% of patients undergoing primary PCI for STEMI have an occasional finding of multivessel coronary artery disease on angiography. In this setting there is a general consensus in the treatment of the culprit lesion (infarct related artery - IRA), while the literature provides contrasting evidence on the preventive treatment of non-culprit coronary lesions (not IRA). Four major randomized trials have, in fact, compared a complete revascularization strategy versus culprit-only revascularization during primary PCI: PRAMI trial, CULPRIT trial, DANAMI-3-PRIMULTI trial and Compare-Acute trial. Although all of these studies demonstrated a benefit in the composite cardiovascular end point in patients undergoing complete revascularization, no statistically significant difference in mortality was found. Therefore, at present, there is no definite evidence on the efficacy of non culprit lesion treatment on mortality and re-MI in patients with STEMI.

The recent guidelines of the European Society of Cardiology 2017 suggest however to evaluate the complete revascularization in multivessel patients before discharge (class IIa, level A). Previous randomized trials such as Compare-Acute study and DANAMI-3-Primulti showed that a complete revascularization strategy guided by FFR, during primary PCI, is associated with a significantly lower risk of cardiovascular events in patients with multivessel disease.

Furthermore, other studies demonstrated that an iFR-guided coronary revascularization is not inferior to FFR-guided revascularization in patients with stable coronary artery disease, whereas, it significantly reduces the overall duration of the procedure. The WAVE study recently demonstrated the diagnostic accuracy of iFR in functional assessment of non-culprit lesions in multivessel patients with STEMI, also highlighting the intralesional reproducibility of both FFR and iFR between baseline and staged. To date, however, there are no studies in the literature that have verified the long-term clinical impact of an iFR-guided revascularization during primary PCI for STEMI patients with multivessel coronary artery disease.

Aim of the study - Multicenter, observational registry to evaluate the long-term clinical impact of an iFR assessment of the non-culprit lesions during primary PCI for STEMI patients with multivessel coronary artery disease.

Methods - patients undergoing primary PCI for STEMI and presenting multivessel disease (at least another coronary stenosis ≥ 50% in addition to the culprit one on QCA analysis) will be enrolled. At the end of the revascularization procedure of the culprit lesion, the functional assessment of the non-culprit lesion will be performed through the use of iFR. In the case of iFR ≤ 0.89, the functionally critical lesion treatment will be performed during the same PCI procedure or staged (at the discretion of the operator and the center). On the other hand, patients with iFR> 0.89 will instead be directed towards a conservative approach with the implementation of clinical-instrumental follow-up.

A clinical follow-up will be performed in all patients by telephone interviews or outpatient visits at 12, 24 and 36 months from the index procedure.

The primary endpoint of the study is represented by the occurrence of Target Lesion Failure (TLF), a composite of cardiovascular death, non-fatal myocardial infarction, and ischemia-driven revascularization of the vessel previously assessed with iFR.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* 12-hour chest pain with ST segment elevation greater than 0.1 mV in at least two contiguous leads treated with primary PCI
* presence of at least one non-culprit lesion with ≥50% stenosis in an epicardial vessel ≥2.5 mm
* informed consent signed

Exclusion Criteria:

* ejection fraction ≤ 30%
* presence of moderate / severe valvulopathies
* electrical instability and hemodynamics at the end of the index procedure (Killip III-IV class)
* TIMI flow <3 at the end of the index procedure
* previous myocardial infarction in the same territory of the non-culprit lesion
* previous coronary artery bypass grafting on the vessel undergoing functional assessment by iFR
* Inability to provide informed consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary PCI for STEMI and presenting with multi vessel coronary disease (at least one ≥ 50% diameter stenosis in a non-infarct-related coronary artery).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  A composite of cardiovascular death, non-fatal myocardial infarction, and ischemia-driven revascularization of the vessel previously assessed with iFR

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Camillo, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided